CLINICAL TRIAL: NCT05450224
Title: Telehealth-delivered Massed Imaginal Exposure for PTSD: Toward Increasing Access to Alternative, Evidence-based Treatment Schedules for Virtual Care
Brief Title: Telehealth-Massed Imaginal Exposure for PTSD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Veteran's Affairs Research and Development Office delays.
Sponsor: Medical University of South Carolina (Other)
Collaborators: Ralph H. Johnson VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00106523
Record Dates: First submitted 2021-11-29; First posted 2022-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Posttraumatic Stress Disorder
Keywords: Veterans
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Telehealth Massed Imaginal Exposure Therapy (Other)
  Interventions: Behavioral: VVC-delivered Massed Imaginal Exposure

INTERVENTIONS:
Behavioral: VVC-delivered Massed Imaginal Exposure — Consistent with Zoellner et al., (2017), six, 60-minute daily sessions of imaginal exposure will be conducted based on the PE manual (Foa et al., 2007). No in vivo exposure or homework will be included. Session 1 will include rationale for imaginal exposure and common reactions to trauma. Sessions 2-6 will focus on imaginal exposure (45 minutes) and processing (15 minutes), with later sessions focused on the most distressing aspect of the trauma memory. The final session will include relapse prevention. All sessions will be delivered within a 10-day window.

SUMMARY:
The purpose of this study is to establish the safety, feasibility, and acceptability of very brief imaginal exposure therapy for post-traumatic stress disorder (PTSD) delivered by telehealth over the course of six-daily 60-minute sessions within a 10-day window. All study visits occur remotely, by telehealth. You will be asked to complete a pre-treatment assessment involving a clinical interview, video-based measures of emotional and physical reactions, such as heart rate and breathing rate, and self-report questionnaires to measure the severity and impact of trauma-related symptoms. These assessments are completed again 1-week, and 1-month after completing treatment. The researchers propose that massed exposure-based therapy delivered via telehealth will advance telemental health treatment options and personalized care for Veterans with PTSD.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65.
* Ability to speak, read, and write English.
* Diagnosis of PTSD based on CAPS-5 (> 3 mo. post-trauma).
* Seeking treatment for PTSD at the Charleston VA.
* Willingness and ability to engage in assessment and treatment visits through VVC, or another VA-approved telehealth videoconferencing platform.

Exclusion Criteria:

* Currently receiving psychotherapy for another anxiety- or stress-related condition.
* Current substance use disorder diagnosis with repeated abuse or dependence within 3 months of study entry and unwillingness to abstain for 24 hours prior to study visits.
* Unstable dose of psychotropic medications within 6 weeks prior to baseline assessment (based on the DMSC; see measures).
* Medical condition that would contraindicate participation in treatment or assessment activities (e.g., severe cardiovascular problems; DMSC, and chart review; see measures).
* Current, or history of bipolar I disorder
* Current, or history of psychotic symptoms
* Serious suicidal risk or a suicide attempt in the past year, as determined by self-report (PHQ-9) and clinical interview (C-SSRS; see measures).
* Active neurological conditions, e.g., seizures, stroke, loss of consciousness or concussion (DMSC, and chart review; see measures)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Adverse events | from admission to 1 month follow up
  Potential adverse events will be assessed with a structured as well as open-ended interview daily during treatment and at follow up.
Satisfaction with treatment - provider | 1 week post-treatment
  PETQ: Prolonged exposure therapist questionnaire; scores range 0-30 with higher scores suggesting patient is more engaged in treatment.
Satisfaction with telehealth - provider | 1 week post-treatment
  TTSQ-Provider: Technology Treatment Satisfaction Questionnaire; scores range 0-30 with higher scores suggesting patient is more engaged in treatment
Satisfaction with treatment - patient | 1 week post-treatment
  STTSR: Satisfaction with Therapy and Therapist Scale-Revised; scores range 0-60 with higher scores indicating higher satisfaction
Satisfaction with telehealth - patient | 1 week post-treatment
  Technology Treatment Satisfaction Questionnaire; scores range 0-60 with higher scores indicating higher satisfaction.
Number of sessions attended per patient | from pre-treatment to 1-month follow-up
  Number of telehealth therapy appointments attended per patient.
Rate of treatment completion and pre-mature dropout. | from pre-treatment to 1-month follow-up
  Total percent of patients retained from initial patients.
CAPS: Clinician-Administered PTSD Scale for DSM-5 | from pre-treatment to 1-month follow-up
  Structured interview for DSM-5 PTSD severity and impairment; Scores range from 0 to 80 with higher scores indicating greater PTSD severity and impairment.
PTSD symptom checklist | from pre-treatment to 1-month follow-up
  PCL-5: PTSD Symptom Checklist for DSM-5. Scores range from 0 to 80, with higher scores indicating greater PTSD severity and impairment.

SECONDARY OUTCOMES:
Remote photoplethysmography | Pre-treatment, 1-week post-treatment, and 1-month follow-up.
  Video-based derivation of psychophysiology including heart rate and respiratory rate
Facial emotional expressivity | Pre-treatment, 1-week post-treatment, and 1-month follow-up.
  Video-based derivation of facial emotional expressivity.
Vocal and linguistic emotional expressivity | Pre-treatment, 1-week post-treatment, and 1-month follow-up.
  Audio-based derivation of vocal and linguistic emotional expressivity.

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-06-28): https://cdn.clinicaltrials.gov/large-docs/24/NCT05450224/Prot_SAP_002.pdf
  • Informed Consent Form (2022-06-07): https://cdn.clinicaltrials.gov/large-docs/24/NCT05450224/ICF_001.pdf